CLINICAL TRIAL: NCT00609440
Title: Morquio's Syndrome: a Case Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated
Sponsor: Clínica de Hidroterapia e Recuperacao Funcional (Other)
Collaborators: Integrated Faculty of Recife (Other)
Responsible Party: Maria do Carmo Pinto Neta, Centro de Hidroterapia e Recuperação Funcional
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mairabelo; MBelo
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-01

CONDITIONS: Morquio's Disease
Keywords: Morquio's disease; physiotherapy; results
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): A single case study, of a patient that was submitted to a physiotherapeutic treatment.
  Interventions: Other: physiotherapeutic treatment

INTERVENTIONS:
Other: physiotherapeutic treatment — At first, the patient was submitted to a conventional physiotherapeutic treatment and respiratory exercises; then, we gave emphasis to the motor development marks and to the march training; eventually, the kid was conducted to hydrotherapy.
  Other Names: physiatry

SUMMARY:
OBJECTIVES: Relating about the benefits proportionated by the physiotherapeutic treatment for the patients that have the Morquio's syndrome. METHODS: This study intends to analyse a patient that presents this syndrome, describing the physiotherapeutic treatment that was proposed and the evolution clinical.

ELIGIBILITY:
Inclusion Criteria:

* The parents agreed with the study;
* The parents signed a consent term

Exclusion Criteria:

* The treatment disturbed the patient physically or emotionally;
* The parents didn't signed the consent term;
* The patient refused to be treated.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-01; Primary Completion 2006-08 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria do Carmo Pinto Neta, Post-graduated, Principal Investigator — Employee